CLINICAL TRIAL: NCT04917250
Title: Gemcitabine, Pegaspargase, Etoposide, and Dexamethasone (GPED) for Patients With Relapsed/Refractory or Advanced NK/T-cell Lymphoma : a Single Arm,Open-lable,Phase II Study
Brief Title: GPED for Patients With Relapsed/Refractory or Advanced NK/T-cell Lymphoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beijing Tongren Hospital (Other)
Responsible Party: Principal Investigator, LIANG WANG, Director of Dept. of Hematology, Beijing Tongren Hospital, Beijing Tongren Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TRhos-ENKTCL-7
Record Dates: First submitted 2021-06-02; First posted 2021-06-08 (Actual); Last update posted 2021-06-08 (Actual); Status verified 2021-06

CONDITIONS: Extranodal NK/T-cell Lymphoma
MeSH Terms: conditions — Lymphoma, Extranodal NK-T-Cell | interventions — Gemcitabine; pegaspargase; Etoposide; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- treatment arm (Experimental): Treated with gemcitabine, pegaspargase, etoposide and dexamethasone
  Interventions: Drug: Gemcitabine; Drug: Pegaspargase; Drug: Etoposide; Drug: Dexamethasone

INTERVENTIONS:
Drug: Gemcitabine — 1000mg/㎡，d1,4 ivdrip
Drug: Pegaspargase — 2500IU/㎡, maximum dose less than 3750IU
Drug: Etoposide — 100mg/㎡，d1-3 ivdrip
Drug: Dexamethasone — 20mg/d d1-4 ivdrip

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of GPED (gemcitabine, pegaspargase, etoposide, and dexamethasone) regimen in the treatment of Relapsed/Refractory or advanced NK/T-cell lymphoma patients

ELIGIBILITY:
Inclusion Criteria:

Histopathology and immunohistochemistry confirmed diagnosis of NK/Tcell lymphoma according to WHO 2016 criteria.

* refractory or relapsed after initial remission, or stage III-IV de novo patients
* PET/CT or CT/MRI with at least one objectively evaluable lesion.
* General status ECOG score 0-3 points.
* The laboratory test within 1 week before enrollment meets the following conditions: Blood routine: Hb>80g/L, PLT>50×10e9/L. Liver function: ALT, AST, TBIL ≤2 times the upper limit of normal. Renal function: Cr is normal. Cardiac function: LVEF≥50%, ECG does not suggest any acute myocardial infarction, arrhythmia or atrioventricular conduction above I Blocking.
* Sign the informed consent form

Exclusion Criteria:

Active infection requires ICU treatment. Concomitant HIV infection or active infection with HBV, HCV. Patients who are infected with HBV but not active hepatitis at the same time are notexcluded.

Significant organ dysfunction Pregnant and lactating women. Had a history of autoimmune diseases, and disease was active in the last 6 months.

Those who were known to be allergic to drugs in the study regimen. Patients with other tumors who require surgery or chemotherapy within 6 months.

• Other experimental drugs are being used.

Ages: 16 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2020-03-20 (Actual); Primary Completion 2021-06-30 (Estimated); Study Completion 2021-08-31 (Estimated)

PRIMARY OUTCOMES:
overall response rate | 24 weeks ±7 days
  evaluated by PET-CT and MRI, according to Lugano 2014 criteria

SECONDARY OUTCOMES:
complete response rate | 24 weeks ±7 days
  evaluated by PET-CT and MRI, according to Lugano 2014 criteria
1-year progression free survival rate | up to 1year after enrollment
  time from date of enrollment to date of disease progression, death of any reason, whichever comes first
1-year overall survival rate | up to 1year after enrollment
  time from date of enrollment to date death of any reason

CONTACTS AND LOCATIONS:
Overall Officials: Liang Wang, M.D., Principal Investigator — Beijing Tongren Hospital
Locations (1):
- Beijing Tongren Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No